CLINICAL TRIAL: NCT05385627
Title: Local Infiltration Analgesia for Foot Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LIA-COHORTE-2022
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Foot surgery; Midfoot surgery; Hindfoot surgery; Forefoot surgery; Ankle surgery; Ankle block; Local infiltration analgesia of the ankle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ankle block: Any participant receiving an ankle block (local infiltration analgesia).
  Interventions: Procedure: Ankle block

INTERVENTIONS:
Procedure: Ankle block — Injection of local anaesthetics at the level of the ankle blindly (local infiltration analgesia). The dose, volume, and type of local anaesthetic will be registered.
  Other Names: Local infiltration analgesia

SUMMARY:
Prospective cohort assessing the effects of ankle block (local infiltration analgesia) on duration of analgesia, pain, opioid consumption, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Surgery of the foot/ankle
* Intraoperative local infiltration analgesia of the ankle
* Age >= 18 years

Exclusion Criteria:

* Inability to read and understand Danish
* Uncooperativeness (judged by investigators)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery of the foot or ankle will be assessed for eligibility. We will attempt to include all adult patients receiving local infiltration analgesia of the ankle for pain management following foot or ankle surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia, measured as time to first pain | 24 hours
  Duration of analgesia measured as time to first pain as reported by the patient. The duration of analgesia is expected to be less than 24 hours. If the duration of analgesia exceeds 24 hours, follow-up will be performed until return of normal sensation is ensured. Duration of analgesia will be set to 24 hours for participants having a duration of analgesia exceeding 24 hours.

SECONDARY OUTCOMES:
Pain in the post-anaesthesia care unit, measured on the Numerical Rating Scale (NRS) | 24 hours
  Pain in the post-anaesthesia care unit as reported by the patient on the NRS (0 to 10 points, 0 no pain, 10 worst perceiveable pain). The assessment will be performed just prior to discharge from the post-anaesthesia care unit.
Participants with failed block | 24 hours
  Failed block will be defined as participants experiencing pain (NRS > 0) prior to discharge from the post-anaesthesia care unit.
Pain at 6 hours postoperatively, measured on the NRS | 6 hours
  Pain at 6 hours postoperatively measured on the NRS as reported by the participant.
Pain at 24 hours postoperatively, measured on the NRS | 24 hours
  Pain at 24 hours postoperatively measured on the NRS as reported by the participant.
Cumulative opioid consumption at 24 hours postoperatively | 24 hours
  Cumulative opioid consumption at 24 hours postoperatively. Opioid consumption will be converted to intravenous morphine equivalents. Intraoperative opioid use will not be included.
Participant satisfaction related to ankle block | 24 hours
  Participants will be asked if they wanted a longer block duration, if they wanted a shorter block duration, and if block duration was adequate (binary outcomes, yes/no).
Unplanned admission | 24 hours
  Most participants will be discharged directly from the post-anaesthesia care unit and some will have planned hospital admission following surgery. Unplanned admission will be defined as an admission that was not planned in advance. The reason for admission will be recorded.
Postoperative nausea and vomiting | 24 hours
  Incidence of postoperative nausea and vomiting.

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Køge, Zealand Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon reasonable request to the coordinating investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available after primary publication with no time limit.
Access Criteria: Reasonable request to the coordinating investigator.